CLINICAL TRIAL: NCT00572325
Title: Concurrent Chemo-radiotherapy for Stage III Non-small Cell Lung Cancer ta an Individualized MLD
Brief Title: Concurrent Chemo-radiation Form NSCLC to a Individualized MLD
Acronym: BRONC CONC MLD
Status: Completed | Type: Observational
Sponsor: Maastricht Radiation Oncology (Other)
Responsible Party: MAASTRO clinic, MAASTRO clinic
Other Study IDs: BRONC CONCURR MLD
Record Dates: First submitted 2007-12-12; First posted 2007-12-13 (Estimated); Last update posted 2010-07-21 (Estimated); Status verified 2010-07

CONDITIONS: Non-small Cell Lung Cancer
Keywords: radiotherapy; NSCLC; stage III non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Inclusion criteria
  * Histological or cytological proven NSCLC
  * UICC stage I-III
  * Performance status 0-2
  * FeV1 and DLCO at least 30% of age-predicted value
  Exclusion criteria:
  * Not NSCLC or mixed NSCLC and other histologies (e.g. small cell carcinoma)
  * stage IV
  * performance status 3 or more
  * FeV 1 or DLCO< 30% of the age-predicted value

SUMMARY:
Our group has shown in a modeling study that increasing the radiation dose to pre-specified normal tissue dose constrains could lead to increased TCP with the same NTCP in patients with non-concurrent chemo-radiation. In a subsequent phase I trial, in patients receiving non-concurrent chemo-radiation we showed the safety of this approach. Here,we want to investigate its efficacy in a prospective study in patients with stage III NSCLC, who are selected for radical concurrent radiotherapy

DETAILED DESCRIPTION:
Eligible patients (see below) will receive radiotherapy to the primary tumor and the initially involved mediastinal lymph nodes to the following MLD (Mean Lung Dose):

* MLD=19 Gy when Fev1 and DLCO>50% of the predicted value
* MLD=15 Gy when Fev1 and/or DLCO 40-49% of the predicted value
* MLD=10 Gy when Fev1 and/or DLCO <40% of the predicted value

Other dose-constrains: spinal cord max: 54 Gy, brachial plexus (Dmax):66 Gy Minimum tumor dose:54 Gy. Maximal tumor dose:69 Gy

Radiotherapy will be delivered as follows:

1. First 3 weeks: 30 fractions: twice-daily fractions of 1.5 Gy, with 8 to 10 h as interfraction-interval, 5 days per week Total dose;45Gy/30 fractions
2. Thereafter: once-daily fractions of 2.0 Gy, 5 days per week until the target dose has been reached.

The radiation doses will be specified according to ICRU 50. Lung density corrections will be applied, as well as all standard QA procedures. Technical requirements are the same as in standard practice at MAASTRO clinic.

Chemotherapy schedules allowed:

1. 1-2 cycles induction chemotherapy; any type will be registered.
2. concurrent part:(day1= first day of radiotherapy)

   1. cisplatin - vinorelbine

      * Cisplatin 50 mg/m2 day 2 and day 9
      * Vinorelbine 20 mg/m2 day 2 and day 9
      * Cisplatin 40mg/m2 day 23
      * Vinorelbine 15mg/m2 day 23 and day 30
   2. cisplatin - docetaxel

      * Cisplatin 50 mg/m2 day 2,9 and 29
      * Docetaxel 20 mg/m2 day 2, 9, 16, 23 and 29
   3. cisplatin - etoposide

      * Cisplatin 60 mg/m2 day 1
      * Docetaxel 120 mg/m2 day 1-3

Q 3 weeks, 3 cycles

When the calculated creatinin clearance is less than 60 ml/min, cisplatin may be substituted for carboplatin

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological proven NSCLC
* UICC stage I-III
* Performance status 0-2
* FeV 1 and DLCO at least 30% of the age-predicted value

Exclusion Criteria:

* Not NSCLC or mixed NSCLC and other histologies (e.g. small cell carcinoma)
* UICC stage IV
* Performance status 3 or more
* FeV 1 and DLCO < 30% of the age-predicted value

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Histological or cytological proven NSCLC
  * UICC stage I-III
  * Performance status 0-2
  * FeV 1 and DLCO at least 30% of the age-predicted value
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2006-08; Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
death | 2,3 and 5 years

SECONDARY OUTCOMES:
-progression-free interval -Dyspnea (CTCAE 3.0) -Dysphagia (CTCAE 3.0) -Patterns of recurrence | 2,3 and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Dirk De Ruysscher, MD,PhD, Principal Investigator — MAASTRO clinic, Maastricht Radiation Oncology
Locations (1):
- MAASTRO clinic, Maastricht Radiation Oncology, Maastricht, Netherlands

REFERENCES:
- [Derived] Nalbantov G, Kietselaer B, Vandecasteele K, Oberije C, Berbee M, Troost E, Dingemans AM, van Baardwijk A, Smits K, Dekker A, Bussink J, De Ruysscher D, Lievens Y, Lambin P. Cardiac comorbidity is an independent risk factor for radiation-induced lung toxicity in lung cancer patients. Radiother Oncol. 2013 Oct;109(1):100-6. doi: 10.1016/j.radonc.2013.08.035. Epub 2013 Sep 14. PMID 24044794
- [Derived] van Baardwijk A, Reymen B, Wanders S, Borger J, Ollers M, Dingemans AM, Bootsma G, Geraedts W, Pitz C, Lunde R, Peters F, Lambin P, De Ruysscher D. Mature results of a phase II trial on individualised accelerated radiotherapy based on normal tissue constraints in concurrent chemo-radiation for stage III non-small cell lung cancer. Eur J Cancer. 2012 Oct;48(15):2339-46. doi: 10.1016/j.ejca.2012.04.014. Epub 2012 May 18. PMID 22608261
- [Derived] Dehing-Oberije C, Aerts H, Yu S, De Ruysscher D, Menheere P, Hilvo M, van der Weide H, Rao B, Lambin P. Development and validation of a prognostic model using blood biomarker information for prediction of survival of non-small-cell lung cancer patients treated with combined chemotherapy and radiation or radiotherapy alone (NCT00181519, NCT00573040, and NCT00572325). Int J Radiat Oncol Biol Phys. 2011 Oct 1;81(2):360-8. doi: 10.1016/j.ijrobp.2010.06.011. Epub 2010 Oct 1. PMID 20888135